CLINICAL TRIAL: NCT04480840
Title: A Randomized, Double-blind, Dose-ranging, Placebo-controlled, Phase 2a Evaluation of the Safety, Tolerability, and Pharmacokinetics of PLN-74809 in Participants With Primary Sclerosing Cholangitis (PSC) and Suspected Liver Fibrosis (INTEGRIS-PSC)
Brief Title: Phase 2a Evaluation of Safety, Tolerability, and Pharmacokinetics of PLN-74809 in Patients With Primary Sclerosing Cholangitis (PSC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pliant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLN-74809-PSC-203; INTEGRIS-PSC (Other: Pliant Therapeutics Inc)
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo (Part 1, 2, and 3)
  Interventions: Drug: Placebo
- PLN-74809 Dose Level 1 (Experimental): Part 1, Cohort 1 Dose: 40 mg, up to 12 weeks
  Interventions: Drug: PLN-74809
- PLN-74809 Dose Level 2 (Experimental): Part 2, Cohort 2 Dose: 80 mg, up to 12 weeks; PLN-74809 Dose Level 2 following PLN-74809 Dose Level 1
  Interventions: Drug: PLN-74809
- PLN-74809 Dose Level 3 (Experimental): Part 2, Cohort 3 Dose: 160 mg, up to 12 weeks; PLN-74809 Dose Level 3 following PLN-74809 Dose Level 1
  Interventions: Drug: PLN-74809
- PLN-74809 Dose Level 4 (Experimental): Part 3, Cohort 4 Dose: 320 mg, for at least 24 weeks and up to 48 weeks; PLN-74809 Dose Level 4 following PLN-74809 Dose Levels 2 and 3
  Interventions: Drug: PLN-74809

INTERVENTIONS:
Drug: PLN-74809 — PLN-74809
  Arms: PLN-74809 Dose Level 1; PLN-74809 Dose Level 2; PLN-74809 Dose Level 3; PLN-74809 Dose Level 4
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Phase 2a, multicenter, randomized, double-blind, dose-ranging, placebo-controlled, study to evaluate the safety, tolerability, and PK of PLN-74809 in participants with primary sclerosing cholangitis and suspected liver fibrosis

DETAILED DESCRIPTION:
Three-part study:

Part 1 - 12-week treatment period evaluating 40 mg of PLN-74809 or matching placebo [Complete] Part 2 - 12-week treatment period evaluating two dose groups, 80 mg and 160 mg of PLN-74809 or matching placebo Part 3 - minimum 24-week, up to 48-week treatment period evaluating 320 mg of PLN-74809 or matching placebo

ELIGIBILITY:
Inclusion Criteria:

* Established clinical diagnosis of large duct PSC based on an abnormal cholangiography as assessed by magnetic resonance cholangiopancreatography (MRCP), endoscopic retrograde cholangiopancreatography (ERCP), and/or percutaneous transhepatic cholangiopancreatography (PTC) in the context of cholestatic liver chemistry
* Suspected liver fibrosis, as defined by liver stiffness measurement (LSM), assessed by ultrasound-based transient elastography (TE, FibroScan®) OR Enhanced Liver Fibrosis (ELF) Score OR Historical liver biopsy showing fibrosis without cirrhosis (by any scoring system) OR Magnetic resonance elastography (MRE)
* Serum ALP concentration within normal limits or > 1 times the upper limit of normal (ULN)
* Participants receiving treatment for IBD are allowed, if on a stable dose from screening and expected to remain stable for the duration of the study
* Serum AST and ALT concentration ≤ 5 times the upper limit of normal
* If receiving treatment with UDCA, therapy is at a dose of < 25 mg/kg/day, has been stable for at least 3 months before screening.

Exclusion Criteria:

* Other causes of liver disease, including secondary sclerosing cholangitis or viral, metabolic, or alcoholic liver disease, as assessed clinically
* Known or suspected overlapping clinical and histologic diagnosis of autoimmune hepatitis
* Small duct PSC with no evidence of large duct involvement (evidence of PSC on historical liver histology, with normal bile ducts on cholangiography)
* Presence of liver cirrhosis as assessed by liver histology, ultrasound-based liver stiffness measurement, ELF score, MRE, and/or signs and symptoms of hepatic decompensation (including but not limited to, jaundice, ascites, variceal hemorrhage, and/or hepatic encephalopathy.
* Serum ALP concentration > 10 times the upper limit of normal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pliant Therapeutics Medical Monitor, Study Director — Pliant Therapeutics, Inc.
Locations (60):
- United States (21):
  - California Liver Research Institute, Pasadena, California
  - Stanford University School of Medicine, Redwood City, California
  - University of California, Davis Medical Center, Sacramento, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - Florida Research Institute, Lakewood Rch, Florida
  - Schiff Center of Liver Diseases/University of Miami, Miami, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital Gastroenterology Liver Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Vanderbilt Digestive Disease Center, Nashville, Tennessee
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
  - VCU Health Clinical Research Services Unit, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Australia (7):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital: Department of Gastroenterology and Hepatology, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred, Melbourne, Victoria
  - St. Vincent's Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Medical University of Vienna Div. of Gastroenterology and Hepatology, Vienna
- Belgium (4):
  - Department Gastroenterology, Hepatopancreatology and Digestive Oncology CUB Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ghent University Hospital, Ghent
  - UZ Leuven, Leuven
- Canada (9):
  - Aspen Woods Clinic, Calgary, Alberta
  - University of Alberta Hospital - Walter C. Mackenzie Health Sciences Centre, Edmonton, Alberta
  - (G.I.R.I) GI Research Institute, Vancouver, British Columbia
  - McMaster University Medical Centre, Hamilton, Ontario
  - London Health Sciences Centre-University Hospital, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto Centre for Liver Disease (TCLD), University Health Network, Toronto General Hospital, Toronto, Ontario
  - Centre de Recherche du Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- France (5):
  - CHU Grenoble Alpes - Hôpital Michallon, Grenoble
  - CHU de Lille service MAD, Lille
  - Saint Antoine Hospital/ Hepatology Department, Paris
  - C.H.U. Hautepierre, Strasbourg
  - Centre Hépato-Biliaire - Hôpital Paul-Brousse, Villejuif
- Germany (5):
  - Charité University Medicine Berlin, Berlin
  - University Hospital Erlangen, Erlangen
  - University Medical Center Hamburg -Eppendorf/ I. Dept of Medicine, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Universitätsmedizin Mainz, I. Med. Klinik, Mainz
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus University Medical Center, Rotterdam
- United Kingdom (4):
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk
  - John Radcliffe Hospital/Oxford University Hospital, Headington, Oxford
  - University Hospitals Birmingham NHS, Birmingham
  - King's College Hospital NHS Foundation Trust, Denmark Hill, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirschfield GM, Kowdley KV, Trivedi PJ, Eksteen B, Hameed B, Vincent C, Chen T, Goel A, Reddy KG, Orman E, Joshi D, Lefebvre EA, Schaub JR, An MC, Clark A, Barnes CN, Pencek R, Thorburn D, Montano-Loza AJ, Schramm C, Bowlus CL, Trauner M, Levy C. Phase II INTEGRIS-PSC trial of bexotegrast, an alphavbeta6/alphavbeta1 integrin inhibitor, in primary sclerosing cholangitis. J Hepatol. 2026 Jan;84(1):86-98. doi: 10.1016/j.jhep.2025.09.016. Epub 2025 Sep 26. PMID 41016442

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: Placebo (Part 1, 2, and 3)
- PLN-74809 Dose Level 1: Part 1, Cohort 1
  Dose: 40 mg, up to 12 weeks
  PLN-74809: PLN-74809
- PLN-74809 Dose Level 2: Part 2, Cohort 2
  Dose: 80 mg, up to 12 weeks; PLN-74809 Dose Level 2 following PLN-74809 Dose Level 1
  PLN-74809: PLN-74809
- PLN-74809 Dose Level 3: Part 2, Cohort 3
  Dose: 160 mg, up to 12 weeks; PLN-74809 Dose Level 3 following PLN-74809 Dose Level 2
  PLN-74809: PLN-74809
- PLN-74809 Dose Level 4: Part 3, Cohort 4
  Dose: 320 mg, for at least 24 weeks and up to 48 weeks; PLN-74809 Dose Level 4 following PLN-74809 Dose Level 3
  PLN-74809: PLN-74809
Period: Overall Study
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Started | 30 | 24 | 20 | 20 | 27
Completed | 28 | 22 | 19 | 19 | 23
Not Completed | 2 | 2 | 1 | 1 | 4
Not completed — Adverse Event | 2 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — illicit drug use | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4 | Total
Number analyzed (Participants) | 30 | 24 | 20 | 20 | 27 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (11.65) | 46.9 (15.06) | 40.5 (15.32) | 45.1 (12.65) | 47.1 (14.47) | 44.9 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 4 | 6 | 14 | 37
  Male | 24 | 17 | 16 | 14 | 13 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 2 | 0 | 7
  Not Hispanic or Latino | 26 | 23 | 18 | 18 | 25 | 110
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 1 | 0 | 7
  White | 25 | 20 | 16 | 18 | 26 | 105
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 10 | 5 | 9 | 9 | 44
  Austria | 1 | 2 | 3 | 1 | 2 | 7
  Netherlands | 1 | 0 | 0 | 0 | 2 | 3
  Belgium | 0 | 0 | 0 | 1 | 1 | 2
  United States | 11 | 12 | 10 | 6 | 4 | 43
  United Kingdom | 3 | 0 | 1 | 3 | 3 | 10
  Australia | 2 | 2 | 0 | 0 | 4 | 8
  France | 1 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 1 | 0 | 2 | 3
BMI at Screening [Mean (Standard Deviation); unit: kg/m^2] | 26.44 (3.562) | 28.21 (5.167) | 26.45 (4.506) | 26.82 (5.950) | 24.60 (3.069) | 26.52 (4.566)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Nature and proportion of TEAEs between PLN-74809 and placebo groups. Treatment-emergent adverse events (TEAEs) are defined as AEs that emerged or worsened in severity after the first administration of study drug
Time Frame: Up to 40 weeks
Population: Safety Population included all participants who took at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 30 | 24 | 20 | 20 | 27
Participants | 21 | 10 | 16 | 15 | 23

2. Primary Outcome: Number of Participants With Serious Treatment Emergent Adverse Events
Description: Nature and proportion of Serious TEAEs between PLN-74809 and placebo groups. An SAE was defined as an event that, at any dose, results in the following: death, a life-threatening situation; in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect or a medically important event or reaction.
Time Frame: Up to 40 weeks
Population: Safety Population included all participants who took at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 30 | 24 | 20 | 20 | 27
Participants | 1 | 1 | 1 | 0 | 1

3. Secondary Outcome: Assessment of PLN-74809 Total Plasma Concentrations at Week 12
Description: Assessment of PLN-74809 Total Plasma Concentrations Week 12, 2 Hour Post Dose
Time Frame: Up to 12 weeks
Population: Pharmacokinetic Population included all participants who took at least 1 dose of study drug with at least one post baseline evaluable PLN-74809 concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PLN-74809 Placebo: Placebo: Placebo (Part 1, 2, and 3)
Arm/Group | PLN-74809 Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 22 | 21 | 18 | 19 | 24
ng/mL | 0.00 (0.00) | 638.71 (378.193) | 843.06 (474.312) | 2035.95 (1020.567) | 3667.50 (1598.067)

4. Secondary Outcome: Assessment of PLN-74809 Total Plasma Concentrations at Week 24
Description: Assessment of PLN-74809 Total Plasma Concentrations Week 24, 2 Hour Post Dose
Time Frame: Up to 24 weeks
Population: Only the dose level 4 and matching placebo cohorts had a treatment period of 24 weeks and were assessed at 24 weeks. Pharmacokinetic Population included all participants who took at least 1 dose of study drug with at least one post baseline evaluable PLN-74809 concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PLN-74809 Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 9 | 0 | 0 | 0 | 22
ng/mL | 0.00 (0.00) |  |  |  | 3583.64 (1642.404)

5. Other Pre Specified Outcome: Assess Change From Baseline in Enhanced Liver Fibrosis (ELF) at Week 12
Description: Enhanced Liver Fibrosis (ELF) score is a non-invasive blood test derived from the measurement of hyaluronic acid (HA), amino terminal propeptide of type III procollagen (PIIINP), and tissue inhibitor of metalloprotease 1 (TIMP1) using a proprietary algorithm (Siemens) which combines the 3 different tests that use 3 different units to produce a number that does not have a unit. ELF score is a laboratory test, is unitless, and is used as a continuous variable. The minimal ELF score is zero, the maximal ELF score is unknown. The higher the ELF score, the worse the disease outcome. ELF is a score of severity assessment against biopsy-proven fibrosis. A score of <7.7 is none to mild, >7.7-9.8 is moderate, >9.8 is severe.
Time Frame: Baseline to week 12
Population: Mean change from baseline in Enhanced Liver Fibrosis Score was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 28 | 21 | 19 | 19 | 26
Unitless | 0.42 (0.75) | 0.16 (0.58) | 0.19 (0.51) | 0.09 (0.55) | 0.19 (0.59)

6. Other Pre Specified Outcome: Assess Change From Baseline in Enhanced Liver Fibrosis (ELF) at Week 24
Description: as for outcome 5
Time Frame: Baseline to week 24
Population: Mean change from baseline in Enhanced Liver Fibrosis Score was assessed in the Full Analysis Set. Only the dose level 4 and matching placebo cohorts had a treatment period of 24 weeks and were assessed at 24 weeks. Participants with baseline and at least one post baseline assessment
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 9 | 0 | 0 | 0 | 24
Unitless | 0.14 (0.58) |  |  |  | 0.19 (0.76)

7. Other Pre Specified Outcome: Assess Change From Baseline in Serum Alkaline Phosphatase (ALP) at Week 12
Description: Liver function Serum Alkaline Phosphatase (ALP) Change from Baseline to Week 12
Time Frame: Baseline to week 12
Population: Participants with baseline and at least one post baseline assessment
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 28 | 22 | 19 | 19 | 25
U/L | 40.2 (130.94) | 7.5 (83.20) | 4.8 (33.56) | -7.5 (34.63) | 1.7 (44.81)

8. Other Pre Specified Outcome: Assess Change From Baseline in Serum Alkaline Phosphatase (ALP) at Week 24
Description: Liver function Serum Alkaline Phosphatase (ALP) Change from Baseline to Week 24
Time Frame: Baseline to week 24
Population: Only the dose level 4 and matching placebo cohorts had a treatment period of 24 weeks and were assessed at 24 weeks. Participants with baseline and at least one post baseline assessment
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 9 | 0 | 0 | 0 | 24
U/L | 34.4 (56.57) |  |  |  | -26.1 (66.55)

9. Other Pre Specified Outcome: Assess Percent Change From Baseline in PRO-C3 Liver Fibrosis Biomarker at Week 12
Description: Assess change in PRO-C3 liver fibrosis biomarker from Baseline to Week 12
Time Frame: Baseline to week 12
Population: Participants with baseline and at least one post baseline assessment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 28 | 21 | 17 | 18 | 25
Percent Change | 22.35 (53.183) | -3.78 (20.471) | 7.12 (20.328) | 5.20 (30.899) | 2.70 (36.130)

10. Other Pre Specified Outcome: Assess Percent Change From Baseline in PRO-C3 Liver Fibrosis Biomarker at Week 24
Description: Assess change in PRO-C3 liver fibrosis biomarker from Baseline to Week 24
Time Frame: Baseline to week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
Number analyzed (Participants) | 9 | 0 | 0 | 0 | 23
Percent Change | -1.38 (36.859) |  |  |  | -12.74 (26.539)

ADVERSE EVENTS:
Time Frame: Up to 40 weeks
Description: All-cause mortality: All Randomized population included all participants who were randomized in the study.
  Adverse Events: Safety population included all participants who took at least 1 dose of study drug.
Arm/Group | Placebo | PLN-74809 Dose Level 1 | PLN-74809 Dose Level 2 | PLN-74809 Dose Level 3 | PLN-74809 Dose Level 4
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/24 | 0/20 | 0/20 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/24 | 1/20 | 0/20 | 1/27
Other Adverse Events (participants affected / at risk) | 21/30 | 10/24 | 16/20 | 15/20 | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | PLN-74809 Dose Level 1 (N=24) | PLN-74809 Dose Level 2 (N=20) | PLN-74809 Dose Level 3 (N=20) | PLN-74809 Dose Level 4 (N=27)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterobacter bacteramia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | PLN-74809 Dose Level 1 (N=24) | PLN-74809 Dose Level 2 (N=20) | PLN-74809 Dose Level 3 (N=20) | PLN-74809 Dose Level 4 (N=27)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 3 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 5 (6)
Fatigue (General disorders) | 5 (6) | 3 (3) | 2 (2) | 4 (5) | 3 (3)
Pyrexia (General disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9) | 2 (2) | 4 (4) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 4 (5) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 4 (6) | 0 (0) | 1 (2) | 1 (1) | 1 (3)
Ocular icterus (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per protocol, the data generated in this clinical study are the exclusive property of the Sponsor and are confidential. Any publication of the results of this study must be authorized by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT04480840/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT04480840/SAP_002.pdf